CLINICAL TRIAL: NCT03221868
Title: Effects of a Physical Exercise Program Among Diabetic Women Users of the National Health System: a Randomized Clinical Trial
Brief Title: Effects of a Physical Exercise Program Among Diabetic Women Users of the National Health System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, MARLOS RODRIGUES DOMINGUES, Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: diabetes7005
Record Dates: First submitted 2016-12-27; First posted 2017-07-19 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus
Keywords: motor activity; women
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical exercise intervention (Experimental): Exercise group. Physical exercise intervention with sessions carried out as circuit-training, three times a week for 12 weeks to improve physical fitness and metabolic control. The sessions will last between 10 and 45 minutes.
  Interventions: Behavioral: Exercise group
- Control (Active Comparator): Control group consisting of women who underwent the same measurements for future comparisons and were assigned to receive information about health and counseling to practice of physical activity.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Exercise group — An exercise-based program following a 12-week periodization using mostly circuit-like activities.
  Arms: Physical exercise intervention
Behavioral: Control group — Counseling to practice physical activity and meetings every 15 days with women to conduct group walks. Booklet with walking schedule and for registering sessions.
  Arms: Control

SUMMARY:
The study aims at evaluating the effects of an intervention among diabetic women (40 years or older) who belong to the Basic Health Units System (Brazilian public health system). The novelty of this project is that the intervention is low cost and demands very little from the health system in terms of structure, facilities and personnel.

DETAILED DESCRIPTION:
The objective of this project is to evaluate the effect of a physical exercise program on the biochemical profile of type 2 diabetic women users of Basic Health Units (BHU) in the urban area of the city of Pelotas (Brazil). This is a randomized clinical trial, where two BHU's of the 14 eligible for the study will be drawn for inclusion in the study. Only those units with more than 100 registered diabetic patients are eligible, they also are not linked to educational institutions and do not present Physical activity projects. Four Basic Health Units (BHU) of the municipality of Pelotas (Brazil) were randomized, two for the intervention group and two for the control group. The intervention group will perform circuit-like physical exercises three times a week and the control will receive counseling to practice physical activity and meetings every 15 days with the womens to carry out walks. The program lasted 12 weeks, with three weekly sessions and presented four distinct sequences containing 10 exercises each, which were performed and circuit form and modified every three weeks. In the first week of the intervention, the women performed a passage in the circuit and with each new week a passage was increased, until the number of three passes was reached (number of passages kept fixed until the end of the intervention). Each exercise initially had a duration of 30 seconds, with a duration of 10 seconds added every three weeks up to a maximum of 60 seconds; The interval of 30 seconds between exercises was kept fixed throughout the intervention. The intensity was controlled by the subjective perception of effort. Mainly blood chemistry will be measured and evaluated.Possible confounding factors to be controlled: age, skin color, schooling, family income, weight, Body Mass Index (BMI), alcohol consumption, smoking, waist circumference, time to diagnose the disease, use of Medicines for diabetes and eating habits. The information will be collected at the baseline, at the eighth week and at the end of the study. Descriptive analyzes of the data will be performed initially, the associations will be tested by correlation, t-test and ANOVA for repeated measures. For comparisons of categorical variables, Chi-square tests will be used for heterogeneity or linear trend. The multivariate analysis will be run through logistic regression. The analyzes will be performed by intention to treat and by adherence, and the level of significance accepted for the study will be 5%. This study will seek to fill gaps in the knowledge about intervention studies in BHU's in order to identify whether physical exercise interventions with proper planning and orientation can promote improvements in the severity of the disease in diabetic women.

ELIGIBILITY:
Inclusion Criteria:

* females;
* type 2 diabetic;
* diagnosed for more than one year;
* BMI ≥25 kg / m²;
* age between 40 and 60 years.

Exclusion Criteria:

* BMI ≥ 40 kg / m²;
* history of stroke;
* neuropathy or severe retinopathy;
* any serious medical condition that prevents the participant to exercise safely;
* history of severe physical disability
* history of acute myocardial infarction in the last six months.

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Measured at baseline, and the end of intervention, 12th week
  - Glycated hemoglobin - %

SECONDARY OUTCOMES:
Change in Glucose | Measured at baseline, and the end of intervention, 12th week
  Fasting glucose - mg/dl
Change in Insulin | Measured at baseline, and the end of intervention, 12th week
  Fasting insulin - μI/ml
Change in BP | Measured at baseline, and the end of intervention, 12th week
  - Blood pressure - mm/hg measured with an automated equipment;
Change in Insulin resistance | Measured at baseline, and the end of intervention, 12th week
  Insulin resistance - Insulin (μI/L) X Fasting Glycemia (mg/dl)/405
Change in Triglycerides | Measured at baseline, and the end of intervention, 12th week
  Triglycerides - mg/dl
Change in Cholesterol | Measured at baseline, and the end of intervention, 12th week
  Total cholesterol and subfractions - mg/dl
Change in CRP | Measured at baseline, and the end of intervention, 12th week
  C-reactive protein - mg/l
Change in CRF | Measured at baseline, and the end of intervention, 12th week
  - Cardiorespiratory fitness - calculated based on the distance covered during the 6-minute walking test;
Change in LLS | Measured at baseline, and the end of intervention, 12th week
  - Lower limb strength - number of repetitions performed during the 30-Second Chair Stand Test;
Change in QoL | Measured at baseline, and the end of intervention, 12th week
  - Quality of life (SF-36) - sum of the scores of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: MARLOS R DOMINGUES, PhD, Principal Investigator — Postgraduate Program in Physical Education, Federal University of Pelotas
Locations (1):
- Physical Education School of the Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No